CLINICAL TRIAL: NCT06175871
Title: Development of a New Clinical Rehabilitation Approach for the Management of Elderly People With a Neuromusculoskeletal Disorder and a Risk of Falls: a Partnership Project Between UQAC and the Specialized Geriatric Services of CIUSSS-SLSJ
Brief Title: New Clinical Rehabilitation Approach for the Management of Falls Risks
Acronym: ReabFalls
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Chicoutimi (Other)
Collaborators: Agence de la Sante et des Services Sociaux du Saguenay-Lac-Saint-Jean (Other)
Responsible Party: Principal Investigator, Rubens da Silva, Director Physical Therapy program, Université du Québec à Chicoutimi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-008
Record Dates: First submitted 2023-11-21; First posted 2023-12-19 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Musculoskeletal Diseases; Chronic Disease; Fall Patients; Aging Problems; Postural Low Back Pain; Parkinson Disease
Keywords: Aging; Rehabilitation; Postural control; Falls; Biomechanics; Technology innovative; Prevention; Mobility
MeSH Terms: conditions — Musculoskeletal Diseases; Chronic Disease; Low Back Pain; Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Clinical trial design
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Otago exercises (Experimental): OTAGO program - based on very specific exercises for balance, force, and muscular endurance as well as on education about the risk of falling. The program is considered as "home care" (exercises to be done at home) but will be done as a group and with supervision, at CIUSSS or from outdoor and nature intervention (recreactional parks). OTAGO session lasts for 30-40 minutes and will be done twice a week at sites with progression. The program is comprised of 5 muscle strengthening exercises and 12 postural balance exercises. Participants will also be invited to walk 2 times per week for 30 minutes (can be divided into shorter periods, for example 3 blocs of 10 minutes) from outdoor sites or recrative parks. According to each person's strength and mobility, exercises will be increased with the use of free weights (for example during squats) and/or by increasing the number of repetitions. Total duration of the program will be 3 months (i.e., a duration adapted to the site).
  Interventions: Other: OTAGO exercises
- Conventional physiotherapy at Hospital (Active Comparator): This group will be for the conventional type of intervention already in place in geriatric services from La Baie Hospital. This therapy used for physiotherapists at site, including mobility exercices.
  Interventions: Other: Conventional therapy

INTERVENTIONS:
Other: OTAGO exercises — Exercices for improvement postural control and mobility and decrease falls risks
  Other Names: plein air et nature exercises
  Arms: Otago exercises
Other: Conventional therapy — Exercice and education from physical therapy practice conventional from Hospital.
  Other Names: Physiotherapy conventional at hospital by clinicians
  Arms: Conventional physiotherapy at Hospital

SUMMARY:
Accidental falls in older adults are one of the world's major pubic health problem, because of their strong association with injuries and mortality rates. In Quebec, falls are responsible for a high rate of hospitalization (more than 1800 emergency department visits every day) and deaths (more than 10,000 in recent years). Preventing falls is therefore a key mission for health professionals. This research program aims to develop a new clinical approach to the rehabilitation management of the older with a neuro-musculoskeletal disorder and a risk of falling. This program is part of a new partnership project between UQAC and specialized geriatric services at the CIUSSS Saguenay-Lac-St-Jean (La Baie site). These geriatric services admit more than 400 new patients per year, representing a large pool of participants for the new program's development. Specifically, this program has 4 phases: 1) Create a clinical profile of patients in rehabilitation care from specialized geriatric services (ex: reasons for consultation, neuro-musculoskeletal disorders, rates and causes of falls, etc.); 2) to diagnose functional deficits of these patients on different dimensions of functional and physical evaluations, using standardized tests and high-tech instruments (ex: platform of force); 3) determine the effectiveness of a new exercise intervention program (OTAGO) for falls prevention; and 4) Measure client and professional team satisfaction as well as long-term impact of this new approach used to prevent falls. The most significant impact of this new program will be to reduce public health expenditure for care of older adults with balance disorder and risk for falls; and therefore, be implanted in other CIUSSS institutions from Quebec.

DETAILED DESCRIPTION:
This research program on aging to create Living Lab Sag aims at maintaining older adult's full individual and collective abilities in the Saguenay-Lac-Saint-Jean (SLSJ) region. The need for innovation and creativity aims at optimizing independence, whether for mobility, the ability to take charge of one's health, to remain at home, to have access to services, and to prevent falls in a frail and aging population. Thus, this program includes expert investigators in the areas of health, engineering and computer science, aging, neuropsychology, geriatrics, and rehabilitation/prevention within a multidisciplinary work approach for durable health for older adults in Saguenay. Living Lab Sag will be implemented based on an enriched research program, approved by the CIUSSS SLSJ (CER# 2019-008) and entitled: Development of a new clinical approach in rehabilitation for the care of older adults with a neuro-musculo-skeletal disorder and a risk of falling: Project in partnership between UQAC and the specialized geriatrics services of the CIUSSS-SLSJ. Canada census reports clearly show the demographic aging of the local population. It is predicted that people 65 years and older will comprise about 24% of the population in 2036, in Canada and Quebec. In parallel with this demographic phenomenon, 50% of Canadians live with at least one chronic disability that is often associated with advanced age, as well as with different neurological, orthopedic and cardiopulmonary degenerative diseases. Some diseases affecting the neuro-musculo-skeletal system will lead to physical disability and to a significant functional limitation in terms of balance, mobility and walking and, consequently, to an increase in the risk of falling. Falls have a significant financial effect on healthcare services. Every year, in Quebec, approximately 1/3 of people aged 65 and over will fall and, sadly, some data suggest that 424,000 people will die, worldwide, because of a fall. The present scenario also shows the importance of developing strategies to reduce the weight of falls on the healthcare system, such as the creation of Living Lab Sag where the older adults will be at the heart of the situation. With team's experience in the area, one strategy among others is the early identification of physical-functional factors leading to a fall, despite the presence of other associated extrinsic factors that are also associated with the fall (i.e., multifactor phenomenon). This identification can be realized through neurophysiological measures from valid and reliable biological signals in rehabilitation, that will help determine the neuromuscular responses associated to the level of physical frailty of the individual and his/her fall risk. However, geriatric services in general don't often have access to high-end screening tools that permit an early detection of balance problems and fall risk. Within an innovative action plan, our research program, in partnership with specialized geriatric services and researchers aims to determine the efficiency of new evaluation and intervention methods for the health of the older adults. Since 2019, this programm integrate new measures using various high-end equipment to capture biological signals enabling to perform research with patients from Hospital and patients from Parkinson Association and community local. The mission of this program is to build a new paradigm for this site while being a reference to evaluate balance/mobility and walking problems, better screen frail older adults who are at risk of falling and direct then to personalized therapy. At this time, this work will develop a longitudinal intervention study using OTAGO (PEO) exercise program. The name "OTAGO" is not an acronym, as "Otago" is a region of New Zealand located southwest of the southern island. PEO is defined by a reeducation program for strength and balance at home (or in a rehabilitation center), that is personalized, and based on conclusive data. The PEO was developed by a geriatrician (Dr. Campbell) and his team of physiotherapists in 1997, after many years of research, to identify the risks of falling and the potential interventions that could reduce these risks. The program exists worldwide but has never been tested in Québec. Although there are different fall prevention programs, conclusive data show the more frequent use of OTAGO because of its efficiency to reduce the risk of death and the incidence rate of falls over a period of one year in an aging population. This program also reduces falls by 25% according to conclusive data, which no other program in Québec and in rural areas has demonstrated until now. Finally, this program can be a cost-effective intervention for the healthcare system by reducing expenses associated to falls in rural areas, and in particular for patients in La Baie Hospital. Already used in Australia and the United States, we have yet to determine its effects in the Saguenay area. The goal is to test and show its efficiency for the fist time in the area by a random clinical trial in La Baie Hospital. This step will make it possible to advance our research program on the effective intervention plan to reduce future public healthcare expenses related to falls. The aim of this study will thus be to evaluate if the PEO, when adapted to La Baie geriatric services, is superior to conventional therapy to improve parameters of walking, balance, muscle activation, postural trunk control, mobility, force, endurance and perception of symptoms related to pain, function, fall risk and, consequently, quality of life (wellbeing), volume of medication and expenses associated to fall. In other step, the purpose is also evaluate the effect of carrying out the OTAGO exercises in an outdoor and nature modality during a feasibility study to see the impact of nature on the functional abilities of older people with neuromusculoskeletal disorders (ex. Parkinson disease).

ELIGIBILITY:
Inclusion Criteria:

* Admitted to La Baie Hospital rehabilitation services; or
* Admitted to the waiting list for geriatric services at La Baie Hospital; or
* Older adults from the communityé
* Age 65 and over
* Able-bodied adult with minimal autonomy to perform fall-prevention tests and exercises.
* Have at least one neuro-musculo-skeletal disorders and risk of falls

Exclusion Criteria:

* Cancer
* Red flags (infection, tumor, etc.)
* Severe psychiatric disorders
* Palliative care
* Congenital spinal deformity (spondylolysis, intervertebral fusions)
* Severe systemic syndromes or diseases that may prevent tests and exercises from being performed.
* Stroke - very acute phase (1 week) and this until medial hemodynamic stability.

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Postural control | change from baseline at 8 to 12 weeks
  Measures of center of pressure (COP) from plateform of force during different balance tasks
Walking | change from baseline at 8 to 12 weeks
  Gait parameters from GaitRite measurement
Trunk postural control on wobble chair | change from baseline at 8 to 12 weeks
  This test measures trunk postural balance during a sitting balance task on an unstable chair where only lumbar spine movements are allowed to restore balance. Briefly, the base of the chair consists of a pivot at its center and four springs that can be arranged and fixed at a distance varying between 6.0 and 21 cm from the center, allowing the system's level of stability to be varied. The system allows only forward/backward and lateral tilting.
Machine learning-driven neuromusculoskeletal (NMS) assessment | change from baseline at 8 to 12 weeks
  Adapt and integrate existing machine learning algorithms (e.g., pose detection, body reconstruction) to create an NMS assessment framework using smartphone cameras. Image and video recording will be done with three smartphone cameras, positioned on tripods at different angles to the participants. The initial use of multiple cameras is crucial for gathering multi-dimensional data and will allow us to evaluate the effect of camera angle, and the number of cameras, on the accuracy and reliability of the analyses. Various scales will be placed within the recording space, serving as reference points for future camera calibration.

SECONDARY OUTCOMES:
Functional mobility test: TUG | change from baseline at 8 to 12 weeks
  To assess mobility. Equipment: A stopwatch. Directions: Patients wear their regular footwear and can use a walking aid, if needed. Begin by having the patient sit back in a standard arm chair and identify a line 3 meters, or 10 feet away, on the floor.
30 Second Sit to Stand Test | change from baseline at 8 to 12 weeks
  The 30CST is a measurement that assesses functional lower extremity strength in older adults. It is part of the Fullerton Functional Fitness Test Battery. This test was developed to overcome the floor effect of the 5 or 10 repetition sit to stand test in older adults.
maximal isometric hand grip strength | change from baseline at 8 to 12 weeks
  Jamar dynamometer to assess maximal isometric hand grip strength and frailty criteria. 3 trials of maximal contraction up 5 seconds. The best value was retained and corrected by body mass index from Fried classification.
Walking test in 10 meters | change from baseline at 8 to 12 weeks
  Walking speed executed in 10 meter walking test. 2 trials and the best value in time seconds was retained for analysis. The Fried criteria by 4,75 meters was also used to measure time in seconds from this distance (14 feet) and normalized by heigth and weigth.
5 times Sit-To-Stand (FTSTS) | change from baseline at 8 to 12 weeks
  If the 30 second sit to stand test was not applied for some patients, we used also this test which it measures the amount of time it takes for a patient to sit and stand five times in succession with arms folded across their chest. 2 trials were applied in this test and the best time in seconds used for analysis.
Numbers of falls | change from baseline at 8 to 12 weeks, 6 and 12 months after
  Self-reported falls before, during and after the study

OTHER OUTCOMES:
Falls Efficacy Scale-International (FES-I) | change from baseline at 8 to 12 weeks
  The Falls Efficacy Scale-International (FES-I) is a short, easy to administer tool that measures the level of concern about falling during social and physical activities inside and outside the home whether or not the person actually does the activity. The level of concern is measured on a four point Likert scale (1=not at all concerned to 4=very concerned).
Pain measures | change from baseline at 8 to 12 weeks
  Pain measurement was applied with the Brain pain inventory (BPI) questionnaire. The interference items were now presented with 0-10 scales, with 0=no interference and 10=interferes completely
Fatigue perception | change from baseline at 8 to 12 weeks
  Fatigue perception used BORG scale during the exercices
Frailty criteria from Fried | change from baseline at 8 to 12 weeks
  The presence of frailty criteria according to Fried was assessed with self-report questions and two physical tests from five characteristics : 1) Low physical activity (to capture history of sedentary behavior or activity: ex. Do you get any physical exercise for the sake of exercising? How often do you leave your house?); 2) fatigue (complaint of exhaustion with normal activity such as walking outside, climbing stairs: ex. I felt that everything I did was an effort in the last week?); 3) weight loss (unintentional weight loss 10 lbs. or more in past year or more than 5% in past year); 4) weakness (grip strength evaluated with manual dynamometer; in average <30 kg for men and <18 kg for women, but data is normalized by body mass index); 5) slowness or slow walking speed (usual gait speed over 4.57 meters (15 feet); ex. >6.5 seconds, dependent of height).
Hoehn and Yahr Scale | Only at baseline from Sample characterization when Parkinson was included.
  The scale has been used for the staging of the functional disability associated with Parkinson's disease.
Cognitive status | Only at baseline from Sample characterization.
  Mini-mental state questionnaire, which was used for grading the cognitive state of patients in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Sharlène Côté, MD, Study Chair — CIUSSS-SLSJ (La Baie Hospital); Julie Bouchard, PhD, Study Director — Université du Québec à Chicoutimi; Patrice Tremblay, PT, Study Chair — CIUSSS-SLSJ (La Baie Hospital); Rubens da Silva, Principal Investigator — Université du Québec à Chicoutimi; Marie-Ève Langelier, MD, Study Chair — Université du Québec à Chicoutimi
Locations (1):
- Rubens da Silva, Saguenay, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fuzhong L, McAuley E, Fisher KJ, Harmer P, Chaumeton N, Wilson NL. Self-efficacy as a mediator between fear of falling and functional ability in the elderly. J Aging Health. 2002 Nov;14(4):452-66. doi: 10.1177/089826402237178. PMID 12391997
- [Background] Poquet N, Lin C. The Brief Pain Inventory (BPI). J Physiother. 2016 Jan;62(1):52. doi: 10.1016/j.jphys.2015.07.001. Epub 2015 Aug 21. No abstract available. PMID 26303366
- [Background] Barry E, Galvin R, Keogh C, Horgan F, Fahey T. Is the Timed Up and Go test a useful predictor of risk of falls in community dwelling older adults: a systematic review and meta-analysis. BMC Geriatr. 2014 Feb 1;14:14. doi: 10.1186/1471-2318-14-14. PMID 24484314
- [Result] Jiang X, Cooper J, Porter MM, Ready AE. Adoption of Canada's Physical Activity Guide and Handbook for Older Adults: impact on functional fitness and energy expenditure. Can J Appl Physiol. 2004 Aug;29(4):395-410. doi: 10.1139/h04-025. PMID 15317981
- [Result] Guideline for the prevention of falls in older persons. American Geriatrics Society, British Geriatrics Society, and American Academy of Orthopaedic Surgeons Panel on Falls Prevention. J Am Geriatr Soc. 2001 May;49(5):664-72. No abstract available. PMID 11380764
- [Result] Woolcott JC, Khan KM, Mitrovic S, Anis AH, Marra CA. The cost of fall related presentations to the ED: a prospective, in-person, patient-tracking analysis of health resource utilization. Osteoporos Int. 2012 May;23(5):1513-9. doi: 10.1007/s00198-011-1764-1. Epub 2011 Sep 3. PMID 21892675
- [Result] Oliveira MR, Vieira ER, Gil AWO, Fernandes KBP, Teixeira DC, Amorim CF, da Silva RA. One-legged stance sway of older adults with and without falls. PLoS One. 2018 Sep 17;13(9):e0203887. doi: 10.1371/journal.pone.0203887. eCollection 2018. PMID 30222769
- [Result] Vieira ER, Tappen R, Gropper SS, Severi MT, Engstrom G, de Oliveira MR, Barbosa AC, da Silva RA. Changes on Walking During Street Crossing Situations and on Dorsiflexion Strength of Older Caribbean Americans After an Exercise Program: A Pilot Study. J Aging Phys Act. 2017 Oct 1;25(4):525-532. doi: 10.1123/japa.2016-0231. Epub 2017 Sep 14. PMID 28095084
- [Result] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Result] Campbell AJ, Robertson MC, Gardner MM, Norton RN, Tilyard MW, Buchner DM. Randomised controlled trial of a general practice programme of home based exercise to prevent falls in elderly women. BMJ. 1997 Oct 25;315(7115):1065-9. doi: 10.1136/bmj.315.7115.1065. PMID 9366737
- [Result] Shubert TE, Smith ML, Goto L, Jiang L, Ory MG. Otago Exercise Program in the United States: Comparison of 2 Implementation Models. Phys Ther. 2017 Feb 1;97(2):187-197. doi: 10.2522/ptj.20160236. PMID 28204770
- [Result] Thomas S, Mackintosh S, Halbert J. Does the 'Otago exercise programme' reduce mortality and falls in older adults?: a systematic review and meta-analysis. Age Ageing. 2010 Nov;39(6):681-7. doi: 10.1093/ageing/afq102. Epub 2010 Sep 4. PMID 20817938
- [Result] Derouesne C, Poitreneau J, Hugonot L, Kalafat M, Dubois B, Laurent B. [Mini-Mental State Examination:a useful method for the evaluation of the cognitive status of patients by the clinician. Consensual French version]. Presse Med. 1999 Jun 12;28(21):1141-8. French. PMID 10399508
- [Result] Jones SE, Kon SS, Canavan JL, Patel MS, Clark AL, Nolan CM, Polkey MI, Man WD. The five-repetition sit-to-stand test as a functional outcome measure in COPD. Thorax. 2013 Nov;68(11):1015-20. doi: 10.1136/thoraxjnl-2013-203576. Epub 2013 Jun 19. PMID 23783372
- [Result] da Silva RA, Vieira ER, Carvalho CE, Oliveira MR, Amorim CF, Neto EN. Age-related differences on low back pain and postural control during one-leg stance: a case-control study. Eur Spine J. 2016 Apr;25(4):1251-7. doi: 10.1007/s00586-015-4255-9. Epub 2015 Oct 1. PMID 26428907
- [Result] Oliveira MR, Vieira ER, Gil AWO, Teixeira DC, Amorim CF, da Silva RA. How many balance task trials are needed to accurately assess postural control measures in older women? J Bodyw Mov Ther. 2019 Jul;23(3):594-597. doi: 10.1016/j.jbmt.2019.04.004. Epub 2019 Apr 12. PMID 31563376
- [Result] Vieira ER, Da Silva RA, Severi MT, Barbosa AC, Amick Iii BC, Zevallos JC, Martinez IL, Chaves PHM. Balance and Gait of Frail, Pre-Frail, and Robust Older Hispanics. Geriatrics (Basel). 2018 Jul 18;3(3):42. doi: 10.3390/geriatrics3030042. PMID 31011080
- [Result] da Silva RA, Vieira ER, Leonard G, Beaulieu LD, Ngomo S, Nowotny AH, Amorim CF. Age- and low back pain-related differences in trunk muscle activation during one-legged stance balance task. Gait Posture. 2019 Mar;69:25-30. doi: 10.1016/j.gaitpost.2019.01.016. Epub 2019 Jan 11. PMID 30658312
- [Result] Dallaire M, Gagnon G, Fortin E, Nepton J, Severn AF, Cote S, Smaili SM, Goncalves de Oliveira Araujo HA, de Oliveira MR, Ngomo S, Bouchard J, da Silva RA. The Impact of Parkinson's Disease on Postural Control in Older People and How Sex can Mediate These Results: A Systematic Review. Geriatrics (Basel). 2021 Oct 29;6(4):105. doi: 10.3390/geriatrics6040105. PMID 34842716
- [Result] de Lima MDCC, Dallaire M, Tremblay C, Nicole A, Fortin E, Maluf IC, Nepton J, Severn AF, Tremblay P, Cote S, Bouchard J, da Silva RA. Physical and Functional Clinical Profile of Older Adults in Specialized Geriatric Rehabilitation Care Services in Saguenay-Quebec: A Retrospective Study at La Baie Hospital. Int J Environ Res Public Health. 2022 Aug 13;19(16):9994. doi: 10.3390/ijerph19169994. PMID 36011629
- See also: Programme d'Exercices OTAGO - Fondation de ma vie - CIUSSS-SLSJ programmes de bourse — https://www.youtube.com/watch?v=AtjiMlHum-4
- See also: Profil main investigator — https://www.uqac.ca/portfolio/rubensdasilva/